CLINICAL TRIAL: NCT00663533
Title: Vasectomy With the Vas-X, a Simple, Minimally Invasive Device for Male Sterilization: A Pilot Study
Brief Title: VAS-2 Vasectomy With the Vax-X
Acronym: VAS-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, John Amory, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 32431-B
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Vasectomy; Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device study only. (No Intervention)
  Interventions: Device: Vas-X

INTERVENTIONS:
Device: Vas-X — mechanical vasectomy device

SUMMARY:
The purpose of this research study is to study an experimental vasectomy device called the Vas-X. This is an experimental study of this new approach to vasectomy.

DETAILED DESCRIPTION:
The Vas-X works by stripping the lining of the vas deferens, the tube that sperm pass through during ejaculation. It is used in a way very similar to routine vasectomy, however, in a routine vasectomy, the vas is burned with an electrical device. With the Vas-X, there is no burning. The investigators are testing the Vas-X to determine whether it will offer a better way of performing a vasectomy.

The investigators will conduct this study at the University of Washington Medical Center, Seattle.

ELIGIBILITY:
Inclusion Criteria:

* healthy male with normal physical findings
* normal testicular volume (15-30mL)
* detectable sperm in ejaculates

Exclusion Criteria:

* Men with past history of

  * hypertension
  * significant cardiovascular
  * thromboembolic disorders
  * renal (including undiagnosed urinary tract bleeding)
  * hepatic, prostatic and testicular disease
  * prior vasectomy or scrotal surgery
  * infertility
* Men with a past history of drug abuse will also be excluded.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
absence of sperm in ejaculated semen 6 months after vasectomy | 6-months

SECONDARY OUTCOMES:
any side effects as well as degree of occlusion of the resected segment of vas deferens | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: John Amory, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Amory JK, Jessen JW, Muller C, Berger RE. Vasectomy by epithelial curettage without suture or cautery: a pilot study in humans. Asian J Androl. 2010 May;12(3):315-21. doi: 10.1038/aja.2009.94. Epub 2010 Feb 15. PMID 20154700